CLINICAL TRIAL: NCT05270603
Title: Comparing the Reliability of a Web-based Intraoperative Adverse Event Assessment Tool With Standard Cognitive Grading. The Intraoperative Complication Assessment and Reporting With Universal Standards - Calculator (ICARUS-C)
Brief Title: The Intraoperative Complication Assessment and Reporting With Universal Standards - Calculator (ICARUS-C)
Acronym: ICARUS-C
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Giovanni Cacciamani, Assistant Professor of Research Urology, University of Southern California
Other Study IDs: UP-21-01010
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Intraoperative Complications; Surgery--Complications; Surgery; Surgical Procedure, Unspecified
Keywords: ICARUS; Intraoperative Complications; ICARUS Calculator
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICARUS Calculator Raters (Intervention Group): Surgeons and anesthesiologists will be asked to use the ICARUS Calculator to grade a subset of 10 clinical scenarios selected from a list of the clinical scenarios and examples from the publications of the 5iAE systems
  Interventions: Other: ICARUS intraoperative adverse events calculator
- Cognitive Grading Raters (Control Group): Surgeons and anesthesiologists will be asked to use the ICARUS Calculator to grade a subset of 10 clinical scenarios (same as the Intervention group) selected from a list of the clinical scenarios and examples from the publications of the 5iAE systems
  Interventions: Other: ICARUS intraoperative adverse events calculator

INTERVENTIONS:
Other: ICARUS intraoperative adverse events calculator — The ICARUS calculator is a web-based tool that uses answers to Boolean, yes/no questions to determine the iAE grade (appendix I). The calculator providers iAE grade outputs for the 5 iAE classification systems.
  https://garnmile.com/iaecalc/
  Development of the ICARUS calculator was performed as follows: Referencing the 5 classification systems, we first assembled a list of Boolean questions based on the iAE grade descriptions. This list was distilled to the minimum number of questions necessary to represent all descriptions in the combined list of iAE grades. Next, these questions were used to independently establish the conditional logic required to determine iAE grade for each classification system. The questions and logic were translated into Hypertext Preprocessor (PHP), a server-side programming language, and JavaScript, a client-side scripting language.

SUMMARY:
As part of the initiative known as the Intraoperative Complication Assessment and Reporting with Universal Standards (ICARUS) project, the investigators are working to develop a set of tools to aid in improving the homogenous reporting of intraoperative adverse events (iAEs). Accordingly, the investigators developed a web-based tool, known as the ICARUS Calculator, that integrates the 5 published iAE grading systems. We plan to compare the consistency of grading responses between the ICARUS Calculator and the individual grading systems as presented in their respective publications.

The purpose of this study is two-fold. First, the investigators hope to evaluate the utility of a web-based intraoperative adverse event (iAE) grading system known as the Intraoperative Complication Assessment and Reporting with Universal Standards (ICARUS) calculator. Second, the investigators plan to evaluate the difference in iAE grading outcomes of the ICARUS calculator compared with standard iAE grading.

DETAILED DESCRIPTION:
Perioperative complications, especially intraoperative adverse events (iAEs), carry significant potential for long-term sequelae in a patient's postoperative course. Without consistent and homogenous reporting, these events represent a substantial gap in contemporary surgical literature and clinical practice. By definition, an iAE is any unplanned incident related to a surgical intervention occurring between skin incision and skin closure. Despite the availability of multiple intraoperative grading and classification systems, colloquiallary known as: EAUiaiC, iAE severity classification scheme, Modified Satava, EAES Grading system, and ClassIntra® (formerly CLASSIC) , the reporting of intraoperative adverse events remains exceedingly rare. Further, while most studies report postoperative adverse events, only a fraction of surgical publications report intraoperative complications as outcomes of interest.

As part of the initiative known as the Intraoperative Complication Assessment and Reporting with Universal Standards (ICARUS) project, the investigators are working to develop a set of tools to aid in improving the homogenous reporting of iAEs. Accordingly, the investigators developed a web-based tool, known as the ICARUS Calculator, that integrates the four aforementioned iAE grading systems. The investigators plan to compare the consistency of grading responses between the ICARUS Calculator and the individual grading systems as presented in their respective publications.

ELIGIBILITY:
Inclusion Criteria:

* Documented understanding, willingness, and agreement to participate in this study
* Males and females; age 18 or older
* Must be either English speaking or fluent with English medical terminology
* Currently or formerly practicing surgeon or proceduralist, regardless of the domain

Exclusion Criteria:

* Activity restrictions that limit one's ability to engage in online survey
* Adults not competent to consent
* Minors, human fetuses, neonates Prisoners/Detainees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study team will identify corresponding authors who have published articles at any point during 2019-2021 in key American and European scientific surgical journals. The study team plans to email up to 1500 authors from each of these journals - though, many of these journals will not likely have substantially fewer corresponding authors. Specifically, these journals will be associated with one or more of the following specialties:
  Anesthesiology Interventional Radiology Interventional Cardiology Cardiothoracic Surgery Colon and rectal surgery General Surgery Gynecologic oncology Gynecology and obstetrics Neurological Surgery Ophthalmologic Surgery Oral and maxillofacial Surgery Orthopaedic Surgery Otorhinolaryngology Plastic Surgery Urology Vascular Surgery
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the consistency and inter-rater reliability of the 5 iAEs grading systems in terms of Distribution of responses by count and percent | 03-01-2022 to 03-15-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Distribution of responses by count and percent
Evaluate the consistency and inter-rater reliability of the 5 iAEs grading systems in terms of Percent agreement of grade | 03-01-2022 to 03-15-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Percent agreement of grade
Evaluate the consistency and inter-rater reliability of the 5 iAEs grading systems using the Cohen's Kappa | 03-01-2022 to 03-15-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  - Cohen's Kappa
Evaluate the consistency and inter-rater reliability of the 5 iAEs grading systems using the Intra-class correlation (ICC) with two-way, random effects to evaluate for consistency of grades | 03-01-2022 to 03-15-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Intra-class correlation (ICC) with two-way, random effects to evaluate for consistency of grades
Evaluate theTime to complete grading (minutes) using the 5 iAEs grading systems | 03-01-2022 to 03-15-2022
  Primary data analysis will involve calculations i to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Time to complete grading (minutes)
Evaluate the consistency and inter-rater reliability of the ICARUS Calculator in term of Distribution of responses by count and percent | 03-16-2022- to 06-01-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Distribution of responses by count and percent
Evaluate the consistency and inter-rater reliability of the ICARUS Calculator in terms of Percent agreement of grade | 03-16-2022- to 06-01-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Percent agreement of grade
Evaluate the consistency and inter-rater reliability of the ICARUS Calculator using Cohen's Kappa | 03-16-2022- to 06-01-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  - Cohen's Kappa
Evaluate the consistency and inter-rater reliability of the ICARUS Calculator using Intra-class correlation (ICC) with two-way, random effects to evaluate for consistency of grades | 03-16-2022- to 06-01-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Intra-class correlation (ICC) with two-way, random effects to evaluate for consistency of grades
Evaluate Time to complete grading (minutes)using the ICARUS Calculator | 03-16-2022- to 06-01-2022
  Primary data analysis will involve calculations to evaluate the consistency and inter-rater agreement for each grading system, as follows:
  -Time to complete grading (minutes)
Determination of benefit in efficiency, consistency, inter-rater reliability of the ICARUS Calculator compared to cognitively grading intraoperative adverse events | 03-16-2022- to 06-01-2022
  Determination of benefit in efficiency, consistency, inter-rater reliability of the ICARUS Calculator compared to cognitively grading intraoperative adverse events
  There will be 5 output groupings involving the grading systems:
  1. ICARUS calculator vs. EAUiaiC
  2. ICARUS calculator vs. iAE severity
  3. ICARUS calculator vs. Modified Satava
  4. ICARUS calculator vs. ClassIntra
  5. ICARUS calculator vs. EAES Classification
Determination of benefit in efficiency of the ICARUS Calculator compared to cognitively grading intraoperative adverse events | 03-16-2022- to 06-01-2022
  Determination of benefit in efficiency, consistency, inter-rater reliability of the ICARUS Calculator compared to cognitively grading intraoperative adverse events
  There will be 5 output groupings involving the grading systems:
  1. ICARUS calculator vs. EAUiaiC
  2. ICARUS calculator vs. iAE severity
  3. ICARUS calculator vs. Modified Satava
  4. ICARUS calculator vs. ClassIntra
  5. ICARUS calculator vs. EAES Classification
Determination of benefit in consistency of the ICARUS Calculator compared to cognitively grading intraoperative adverse events | 03-16-2022- to 06-01-2022
  Determination of benefit in efficiency, consistency, inter-rater reliability of the ICARUS Calculator compared to cognitively grading intraoperative adverse events
  There will be 5 output groupings involving the grading systems:
  1. ICARUS calculator vs. EAUiaiC
  2. ICARUS calculator vs. iAE severity
  3. ICARUS calculator vs. Modified Satava
  4. ICARUS calculator vs. ClassIntra
  5. ICARUS calculator vs. EAES Classification
Determination of benefit in inter-rater reliability of the ICARUS Calculator compared to cognitively grading intraoperative adverse events | 03-16-2022- to 06-01-2022
  Determination of benefit in efficiency, consistency, inter-rater reliability of the ICARUS Calculator compared to cognitively grading intraoperative adverse events
  There will be 5 output groupings involving the grading systems:
  1. ICARUS calculator vs. EAUiaiC
  2. ICARUS calculator vs. iAE severity
  3. ICARUS calculator vs. Modified Satava
  4. ICARUS calculator vs. ClassIntra
  5. ICARUS calculator vs. EAES Classification

SECONDARY OUTCOMES:
Evaluation of the experience using the ICARUS calculator by System Usability Scale (SUS) questionnaire | 03-16-2022- to 06-01-2022
  Assess the physician satisfaction using a validated questionnaires System Usability Scale (SUS) questionnaire
Evaluation of the experience using the ICARUS calculator by using the Usefulness, Satisfaction and Ease of Use (USE) questionnaire. | 03-16-2022- to 06-01-2022
  Assess the physician satisfaction using a validated questionnaires: Questionnaire for User Interaction Satisfaction (QUIS) and Usefulness, Satisfaction and Ease of Use (USE) questionnaire
Evaluation of the experience using the ICARUS calculator by using Questionnaire for User Interaction Satisfaction (QUIS) | 03-16-2022- to 06-01-2022
  Assess the physician satisfaction using a validated questionnaires: Questionnaire for User Interaction Satisfaction (QUIS)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cacciamani, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biyani CS, Pecanka J, Roupret M, Jensen JB, Mitropoulos D. Intraoperative Adverse Incident Classification (EAUiaiC) by the European Association of Urology ad hoc Complications Guidelines Panel. Eur Urol. 2020 May;77(5):601-610. doi: 10.1016/j.eururo.2019.11.015. Epub 2019 Nov 29. PMID 31787430
- [Background] Kaafarani HM, Mavros MN, Hwabejire J, Fagenholz P, Yeh DD, Demoya M, King DR, Alam HB, Chang Y, Hutter M, Antonelli D, Gervasini A, Velmahos GC. Derivation and validation of a novel severity classification for intraoperative adverse events. J Am Coll Surg. 2014 Jun;218(6):1120-8. doi: 10.1016/j.jamcollsurg.2013.12.060. Epub 2014 Feb 28. PMID 24702887
- [Background] Kazaryan AM, Rosok BI, Edwin B. Morbidity assessment in surgery: refinement proposal based on a concept of perioperative adverse events. ISRN Surg. 2013 May 16;2013:625093. doi: 10.1155/2013/625093. Print 2013. PMID 23762627
- [Background] Dell-Kuster S, Gomes NV, Gawria L, Aghlmandi S, Aduse-Poku M, Bissett I, Blanc C, Brandt C, Ten Broek RB, Bruppacher HR, Clancy C, Delrio P, Espin E, Galanos-Demiris K, Gecim IE, Ghaffari S, Gie O, Goebel B, Hahnloser D, Herbst F, Ioannidis O, Joller S, Kang S, Martin R, Mayr J, Meier S, Murugesan J, Nally D, Ozcelik M, Pace U, Passeri M, Rabanser S, Ranter B, Rega D, Ridgway PF, Rosman C, Schmid R, Schumacher P, Solis-Pena A, Villarino L, Vrochides D, Engel A, O'Grady G, Loveday B, Steiner LA, Van Goor H, Bucher HC, Clavien PA, Kirchhoff P, Rosenthal R. Prospective validation of classification of intraoperative adverse events (ClassIntra): international, multicentre cohort study. BMJ. 2020 Aug 25;370:m2917. doi: 10.1136/bmj.m2917. PMID 32843333
- [Background] Francis NK, Curtis NJ, Conti JA, Foster JD, Bonjer HJ, Hanna GB; EAES committees. EAES classification of intraoperative adverse events in laparoscopic surgery. Surg Endosc. 2018 Sep;32(9):3822-3829. doi: 10.1007/s00464-018-6108-1. Epub 2018 Feb 12. PMID 29435754
- [Background] Cacciamani G, Sholklapper T, Sotelo R, Desai M, Gill I. A Protocol for the Development of the Intraoperative Complications Assessment and Reporting With Universal Standards Criteria: The ICARUS Project. Int J Surg Protoc. 2021 Aug 6;25(1):160-164. doi: 10.29337/ijsp.155. eCollection 2021. PMID 34430764